CLINICAL TRIAL: NCT05652270
Title: Maximizing Patient Goal Attainment, Motivations and Expectations (mGAME) in Elective Musculoskeletal Care
Brief Title: Maximizing Patient Goal Attainment
Acronym: mGAME
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Medacta USA (Industry)
Responsible Party: Principal Investigator, Kevin.J.McGuire, Section Chief for Center for Pain and Spine, Assistant Professor of Orthopaedics, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY02001760
Record Dates: First submitted 2022-12-07; First posted 2022-12-15 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2024-12

CONDITIONS: Knee Osteoarthritis; Knee Injuries; Knee Pain Chronic; Knee Injuries and Disorders
Keywords: Orthopaedic; Knee; Patient Goals
MeSH Terms: conditions — Osteoarthritis, Knee; Knee Injuries; Disease | interventions — Sustainable Development

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Goal Attainment Intervention (Active Comparator)
  Interventions: Behavioral: Goal Attainment
- Goal Development Intervention (Active Comparator)
  Interventions: Behavioral: Goal Development
- Goal Development and Tracking Intervention (Active Comparator)
  Interventions: Behavioral: Goal Development; Behavioral: Goal Tracking

INTERVENTIONS:
Behavioral: Goal Attainment — Development of an attainable goal
  Arms: Goal Attainment Intervention
Behavioral: Goal Development — A Systematic process to help patients create "SMaRT " goals
  Arms: Goal Development Intervention; Goal Development and Tracking Intervention
Behavioral: Goal Tracking — Setting milestones to allow patients to track their progress towards their developed goal
  Arms: Goal Development and Tracking Intervention

SUMMARY:
To evaluate the effectiveness of the goal development intervention in guiding individual patients through the identification of high quality, specific, measurable, relevant and time-bound goal for treatment.

ELIGIBILITY:
Inclusion Criteria:

* Individuals 21 years of age or older
* New patients or existing patients with a new problem that are scheduled to see an orthopaedic surgeon in the Hip and Knee Arthroplasty service for a knee consult.

Exclusion Criteria:

* Individuals who are unable to consent or complete surveys without assistance
* Non-English speaking
* Patients who are less than 12 months from surgery on the knee they are being evaluated for, less than 6 months from surgery on the spine, or less than 3 months from another knee/hip surgery

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2023-04-21 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effectiveness of the goal development intervention using the Goal Attainment Outcome Measure | 8 Months
  To evaluate the effectiveness of the goal development intervention in guiding individual patients through the identification of high quality, specific, measurable, relevant and time-bound goal for treatment.

SECONDARY OUTCOMES:
To assess the intervention's ability to improve shared decision making using the collaboRATE measure | 8 Months
  To assess the acceptability, usability, as well as qualitatively the appropriateness, feasibility, and scalability of integrating the brief patient goal development intervention into standard clinical care. To assess the intervention's ability to improve shared decision making.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin J McGuire, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No